CLINICAL TRIAL: NCT00538993
Title: Improving Provider Counseling Interventions in HIV Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H97HA01144
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Provider receives cue sheet to assist with counseling.
  Interventions: Behavioral: Stage based counseling
- 2 (No Intervention): Provider does not receive cue sheet.

INTERVENTIONS:
Behavioral: Stage based counseling
  Arms: 1

SUMMARY:
Hypothesis: HIV clinicians trained to deliver brief counseling messages and receiving cues from a brief computer survey on risk behaviors of their patients can counsel have an impact on patient's risk behaviors.

DETAILED DESCRIPTION:
This is a randomized controlled study. The purpose of this study is to assess the impact of the cue sheet as an aid to targeted provider behavioral counseling. All enrolled participants are HIV+ adults seen for regular medical care at a site affiliated with the Johns Hopkins AIDS Service. After consenting, participants will take an audio-assisted computer interviews to collect patient risk assessment data. For participants randomized to the intervention arm, the printed output on risk behaviors is then given to the provider along with cues for staged-based counseling for use during the same visit. Participants in the control arm take the same computerized risk assessment but there are no printed cue sheets. Risk behaviors of all participants are assessed at entry, at 6 months, and at 12 months. The main outcome measure is change in HIV transmission behaviors at 12 months for those in the intervention arm compared to the control arm.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive
* English speaking

Exclusion Criteria:

* Cannot give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2003-09 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Disclosure of HIV status to sex partners; unprotected sexual encounters. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Emily Erbelding, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States